CLINICAL TRIAL: NCT02126748
Title: The Effectiveness of Assisted Autogenic Drainage (AAD) and Intrapulmonary Percussive Ventilation (IPV) to Treat Hospitalized Infants (<2years) With Acute Viral Bronchiolitis: a Randomised Clinical Trial.
Brief Title: The Effectiveness of AAD and IPV to Treat Hospitalized Infants (<2years) With Acute Viral Bronchiolitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Filip Van Ginderdeuren, PT,Drs, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FVG003
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; Wang score; Sa02; airway clearance techniques; intrapulmonary percussive ventilation; assisted autogenic drainage
MeSH Terms: conditions — Bronchiolitis | interventions — Inhalation; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intrapulmonary Percussive Ventilation (Experimental): 20 min of IPV administered to the patient inhalation 4ml hypertonic saline 3% 3x/day
  Interventions: Other: inhalation 4ml hypertonic saline 3% 3x/day; Device: Intrapulmonary Percussive Ventilation
- Assisted Autogenic Drainage (Active Comparator): 20 min of AAD administered to the patient inhalation 4ml hypertonic saline 3% 3x/day
  Interventions: Other: inhalation 4ml hypertonic saline 3% 3x/day; Procedure: Assisted Autogenic Drainage
- control (No Intervention): 20 min of bouncing administered tot the patient inhalation 4ml hypertonic saline 3% 3x/day

INTERVENTIONS:
Other: inhalation 4ml hypertonic saline 3% 3x/day
  Arms: Assisted Autogenic Drainage; Intrapulmonary Percussive Ventilation
Device: Intrapulmonary Percussive Ventilation
  Arms: Intrapulmonary Percussive Ventilation
Procedure: Assisted Autogenic Drainage
  Arms: Assisted Autogenic Drainage

SUMMARY:
The purpose of this study is to investigate the effectiveness of two airway clearance techniques; Intrapulmonary Percussive Ventilation and Assisted Autogenic Drainage in hospitalized infants under the age of 2 with acute viral bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* first period of wheezing
* Wang score between 3 and 7
* age < 24 months
* Sa02> 90%

Exclusion Criteria:

* ICU patients
* mechanical ventilation
* use of antibiotics
* use of corticosteroids
* gestational age < 34 weeks
* chronic cardiac or pulmonary disease
* no parental consent

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Uz Brussel, Jette, Brussels Capital, Belgium

REFERENCES:
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196

RESULTS

PARTICIPANT FLOW:
Groups:
- Intrapulmonary Percussive Ventilation: 20 min of IPV administered to the patient inhalation 4ml hypertonic saline 3% 3x/day
  inhalation 4ml hypertonic saline 3% 3x/day
  Intrapulmonary Percussive Ventilation
- Assisted Autogenic Drainage: 20 min of AAD administered to the patient inhalation 4ml hypertonic saline 3% 3x/day
  inhalation 4ml hypertonic saline 3% 3x/day
  Assisted Autogenic Drainage
- Control: 20 min of bouncing administered to the patient inhalation 4ml hypertonic saline 3% 3x/day
Period: Overall Study
Arm/Group | Intrapulmonary Percussive Ventilation | Assisted Autogenic Drainage | Control
Started | 33 | 34 | 36
Completed | 31 | 31 | 31
Not Completed | 2 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrapulmonary Percussive Ventilation | Assisted Autogenic Drainage | Control | Total
Number analyzed (Participants) | 31 | 31 | 31 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 31 | 31 | 93
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 18 | 49
  Male | 16 | 15 | 13 | 44
Region of Enrollment [Number; unit: participants]
  Belgium | 31 | 31 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Previously publised data ( Luo et al. 2011) showed that the average hospital stay for infants with acute viral bronchiolitis, inhaling 4 ml NaCl3%, three times /day is 6 days ( SD 1,2)
Time Frame: 6 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intrapulmonary Percussive Ventilation | Assisted Autogenic Drainage | Control
Number analyzed (Participants) | 31 | 31 | 31
days | 3.5 (1.3) | 3.6 (1.4) | 4.5 (1.9)

2. Secondary Outcome: Wang Score
Time Frame: before treatment, immediately after treatment and 1h after treatment
Reporting Status: Not Posted

3. Secondary Outcome: Heartrate
Time Frame: before, after and 1h after intervention
Reporting Status: Not Posted

4. Secondary Outcome: Oxygen Saturation (SaO2)
Description: oxygen saturation (SaO2) measured by pulse -oximetry
Time Frame: before, after and 1h after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intrapulmonary Percussive Ventilation | Assisted Autogenic Drainage | Control
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No